CLINICAL TRIAL: NCT00801450
Title: Intravitreal Injection Versus Sub-Tenon's Infusion of Triamcinolone Acetonide for Refractory Diabetic Macular Edema During Cataract Surgery
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Rodrigo Jorge, University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2995/2007
Record Dates: First submitted 2008-12-02; First posted 2008-12-03 (Estimated); Last update posted 2009-10-12 (Estimated); Status verified 2009-10

CONDITIONS: Diabetic Macular Edema
Keywords: diabetes; macular edema; triamcinolone; cataract; refractory diabetic macular edema
MeSH Terms: conditions — Diabetes Mellitus; Macular Edema; Cataract | interventions — Triamcinolone Acetonide

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intravitreal (IVI) (Experimental)
  Interventions: Drug: Triamcinolone acetonide
- SubTenon´s (STI) (Experimental)
  Interventions: Drug: Triamcinolone acetonide

INTERVENTIONS:
Drug: Triamcinolone acetonide — 4 mg
  Arms: Intravitreal (IVI)
Drug: Triamcinolone acetonide — 40 mg
  Arms: SubTenon´s (STI)

SUMMARY:
Triamcinolone has already been used by different routes of administration to treat diabetic macular edema. In the present study, intravitreal injection (IVI) and posterior sub-Tenon's infusion (STI) of triamcinolone acetonide (TA) during phacoemulsification cataract surgery in eyes with refractory diffuse diabetic macular edema are tested.

ELIGIBILITY:
Inclusion Criteria:

* Refractory diffuse DME unresponsive to focal laser photocoagulation
* Best corrected visual acuity between 20/800 and 20/40; Central subfield macular thickness greater than 300 µm

Exclusion Criteria:

* Previous ocular surgery
* Glycosylated hemoglobin (Hb A1C) rate above 10%
* History of glaucoma or ocular hypertension
* Loss of vision as a result of other causes
* Systemic corticoid therapy
* Severe systemic disease
* Any condition affecting follow-up or documentation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2007-09; Primary Completion 2008-12 (Estimated); Study Completion 2009-02 (Estimated)

PRIMARY OUTCOMES:
central subfield macular thickness | baseline and at 2, 4, 8±1 ,12±2 and 24±2 weeks postoperatively

SECONDARY OUTCOMES:
Best Corrected Visual Acuity | baseline and at 2, 4, 8±1, 12±2 and 24±2 weeks postoperatively
Intraocular pressure | baseline and at 2, 4, 8±1 ,12±2 and 24±2 weeks postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital das Clínicas da Faculdade de Medicina de Ribeirão Preto da Universidade de São Paulo, Ribeirão Preto, São Paulo, Brazil

REFERENCES:
- [Background] Kumar V, Ghosh B, Raina UK, Goel N. Comparative therapy evaluation of intravitreal bevacizumab and triamcinolone acetonide on persistent diffuse diabetic macular edema. Am J Ophthalmol. 2008 Dec;146(6):974; author reply 974-5. doi: 10.1016/j.ajo.2008.08.013. No abstract available. PMID 19027427
- [Background] Audren F, Lecleire-Collet A, Erginay A, Haouchine B, Benosman R, Bergmann JF, Gaudric A, Massin P. Intravitreal triamcinolone acetonide for diffuse diabetic macular edema: phase 2 trial comparing 4 mg vs 2 mg. Am J Ophthalmol. 2006 Nov;142(5):794-99. doi: 10.1016/j.ajo.2006.06.011. Epub 2006 Sep 15. PMID 16978576
- [Background] Bonini-Filho MA, Jorge R, Barbosa JC, Calucci D, Cardillo JA, Costa RA. Intravitreal injection versus sub-Tenon's infusion of triamcinolone acetonide for refractory diabetic macular edema: a randomized clinical trial. Invest Ophthalmol Vis Sci. 2005 Oct;46(10):3845-9. doi: 10.1167/iovs.05-0297. PMID 16186372
- [Background] Paccola L, Costa RA, Folgosa MS, Barbosa JC, Scott IU, Jorge R. Intravitreal triamcinolone versus bevacizumab for treatment of refractory diabetic macular oedema (IBEME study). Br J Ophthalmol. 2008 Jan;92(1):76-80. doi: 10.1136/bjo.2007.129122. Epub 2007 Oct 26. PMID 17965109